CLINICAL TRIAL: NCT03852004
Title: Comparison of Osteopathic Treatment Versus Simulation on Motor Development of Hypotonic Infants.
Brief Title: Osteopathic Treatment on Motor Development of Hypotonic Infants.
Acronym: HYPOSTEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Collaborators: Centre Broussais (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HYPOSTEO
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Hypotonia
Keywords: osteopathy; hypotonia; children
MeSH Terms: conditions — Muscle Hypotonia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: simulated osteopathic treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopatic treatment (Experimental): An osteopatic treatment will be realised by osteopath
  Interventions: Other: ostheopathy
- simulated osteopathic treatment (Placebo Comparator): A simulated ostepathic treatment will be realised by osteopath
  Interventions: Other: simulated osteopathic treatment

INTERVENTIONS:
Other: ostheopathy — standardized osteopathic treatment
  Arms: Osteopatic treatment
Other: simulated osteopathic treatment — standardized simulated osteopathic treatment
  Arms: simulated osteopathic treatment

SUMMARY:
Interventional study involving the human at risk and minimal constraint (RIPH2), randomized single-blind comparing the impact of osteopathic treatment on the axial tone of the hypotonic infant versus simulation

DETAILED DESCRIPTION:
Children referred to the "Center Broussais" clinic for hypotonia are evaluated in terms of psychomotor development by a pediatrician competent in neuro-pediatrics. It is a cabinet for the care of children from 0 to 16 years.

Osteopaths and pediatricians work together in this office of which 50% are children with neurological disorders.

If osteopathic care is indicated, and for children with inclusion / non-inclusion criteria, the study will be offered to parents. In case of parental acceptance, children will be randomized in single blind to receive either an osteopathic treatment (osteo group) or a simulation (simulation group). Neither the parents nor the pediatrician will know the randomization group.

The osteopathic treatment or simulation will be performed in a standardized way according to a previously established protocol.

In both groups, a neurological evaluation of the axial tone will be performed by a pediatrician before randomization, at the end of the first consultation and at the end of the 3rd consultation, ie 3 consultations by a pediatrician.

If the child was drawn in the "simulation" group, three additional consultations will be offered at the end of the study to allow him to benefit from optimal osteopathic care

ELIGIBILITY:
Inclusion Criteria:Age: 8 months-24 months corrected age Axial hypotonia in the neurological examination

* Age (age corrected for prematurity) of motor development evaluated on the Denver II scale below chronological age
* Proposal for osteopathic treatment by the pediatrician or treating physician

Exclusion Criteria:

* • Fever, shock or recent fall (face, skull, spine) not medically investigated, persistent cyanosis, bulging or depressed fontanel, cervical stiffness, fever

  * Neuromuscular diseases without axial hypotonia
  * Not affiliated to a social security scheme
  * Refusal to participate in the study by parents

Ages: 8 Months to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2025-06-13 (Estimated); Study Completion 2026-01-13 (Estimated)

PRIMARY OUTCOMES:
Motor development on the Denver II scale | at month 6
  Comparison of the difference between chronological age (in corrected age) and motor development age on the Denver II motor scale in the 2 groups after 3 osteopathy consultations or simulation

SECONDARY OUTCOMES:
Motor development on the Denver II scale | at month 2
Motor development on the Denver II scale | at month 4
Satisfaction visual scale (from 0 to 10) | at month 6
  comparison of parents satisfaction with a visual analogic scale in the 2 groups

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHI Creteil, Créteil
  - Centre Broussais, Paris

IPD SHARING:
Plan to Share IPD: No